CLINICAL TRIAL: NCT04710342
Title: A Non-Randomized Clinical Study Evaluating Use of the CapBuster Medical Device System for the Crossing of Chronic Total Occlusions
Brief Title: Clinical Study Evaluating Use of the CapBuster Medical Device System for the Crossing of Chronic Total Occlusions
Acronym: CapBuster
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Praxis Medical Devices Ltd (Industry)
Collaborators: Ospedale Regionale di Lugano (Other); St. Antonius Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAP0001
Record Dates: First submitted 2021-01-11; First posted 2021-01-14 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Chronic Total Occlusion

STUDY DESIGN:
Intervention Model Description: If crossing the CTO is not successful with a conventional guidewire, the CapBuster system will be used to try to cross the occlusion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CTO proximal cap crossing (Experimental): To demonstrate that CapBuster breaks the proximal cap of CTO's
  Interventions: Device: CapBuster

INTERVENTIONS:
Device: CapBuster — Evaluate the safety and effectiveness of the CapBuster System in crossing de novo or restenotic chronic total occlusions in infrapopliteal peripheral arteries.

SUMMARY:
This study represents a prospective, non-randomized, dual-center clinical study to evaluate the safety and effectiveness of the CapBuster System in crossing a de novo or restenotic infrapopliteal chronic total occlusion.

Measures of safety and efficacy will be assessed through 30 days post-intervention.

DETAILED DESCRIPTION:
The diagnostic and interventional procedure can be conducted via contralateral or antegrade approach and arterial access will be obtained utilizing standard percutaneous techniques and devices. Baseline angiographic images will be obtained prior to the study intervention to confirm the presence of a peripheral arterial occlusion. These images will include the target lesion as well as inflow and outflow with ipsilateral run off to the distal foot. If angiographic imaging confirms that the subject meets enrollment criteria, the enrolled subject will then undergo the study procedure.

If the investigator determines that treatment is required of non-target arterial lesions, the treatment may be performed during the study index procedure according to the investigator's standard practices using commercially available devices.

Prior to utilization of the CapBuster system, the investigator will attempt to cross the target lesion CTO utilizing conventional catheters and guidewires. To minimize vessel trauma, attempted guidewire crossing time will be limited to no more than 5 minutes. The crossing time will begin when the guidewire reaches the lesion CTO cap and will end after occlusion is successfully crossed with confirmed wire placement in the true lumen. If successful crossing is achieved with a conventional guidewire, the CapBuster system will not be utilized. The subject will be a screen failure and will not be considered enrolled in the trial.

If crossing attempt is not successful with a conventional guidewire, the CapBuster system will be utilized. A subject is considered enrolled in the study upon introduction of the CapBuster system into the subject's vasculature. The CapBuster support catheter will be inserted over a conventional guidewire and advanced until the distal tip reaches the CTO cap. The CapBuster 3.0 mm diameter balloon is then inflated to stabilize the system within the arterial vessel. The conventional guidewire is replaced with the CapBuster penetrating wire and, under fluoroscopic guidance, the penetrating wire is manually rotated to penetrate the CTO cap. The balloon pressure may be increased to ensure proper apposition with the vessel wall and maximize stability. Following penetration of the cap, the penetrating wire is replaced with a conventional steerable guidewire. Standard wire escalation techniques will be utilized for continued advancement of the conventional guidewire and complete crossing of the occlusion.

Angiography is performed to confirm guidewire placement. Successful crossing is defined as guidewire placement within the true lumen proximal and distal to the target lesion without utilization of a re-entry device.

After successful crossing is achieved, the target lesion may be treated per Investigator discretion with commercially available devices.

ELIGIBILITY:
Inclusion Criteria:

1. Males > 18 years of age and Female patients of non child-bearing potential
2. Clinical diagnosis of peripheral arterial disease requiring revascularization as evidenced by Duplex UltraSound, Digital Subtraction Angiography, CT angiography, or MR angiography
3. Rutherford Classification 2-5
4. Presence of infrapopliteal arterial de novo or restenotic chronic total occlusion(s) (100% stenosis), with TIMI 0 flow, confirmed by angiography. Vessel distal to the occlusion(s) must be visualized per collateral or retrograde flow. A maximum of 2 target occlusions can be treated per patient. Target occlusion(s) can be in-stent restenosis
5. Target vessel(s) must be ≥ 2.5 mm and ≤ 3.25 mm in diameter proximal to the target occlusion(s) by visual estimate
6. Target occlusions(s) cannot be crossed by conventional guidewire (crossing time limited to ≤5 minutes)
7. In the opinion of the investigator, life expectancy of > 1 year
8. Willing and able to sign the informed consent form

Exclusion Criteria:

1. Target occlusion is within a bypass graft
2. Target occlusion can be crossed by conventional guidewire
3. Target occlusion is below tibiotalar joint
4. Presence of acute limb ischemia
5. Known sensitivity or allergy to contrast materials that cannot be adequately pre-treated
6. Known allergy or contraindication to all antiplatelet therapy
7. Subject has signs or symptoms of systemic infection/sepsis (temperature ≥38.0o Celsius and WBC ≥12,000 cells/uL). If subject has localized infection, including cellulitis or osteomyelitis, or infection is adequately treated and controlled, per investigator discretion, patient may be enrolled.
8. Known or suspected myocardial infarction or stroke within previous 30 days
9. Significant acute or chronic renal disease with a GFR <30 mL/min/1.73m2
10. History of a surgical or endovascular procedure on the target limb within 30 days of the index procedure or non-target limb within 2 weeks of the index procedure
11. Planned surgical or endovascular procedure prior to the subject's 30-day follow-up. Planned minor amputations are allowed.
12. Subject is scheduled for a target limb major amputation (above the ankle) within 30 days post study procedure
13. Currently participating in another investigational drug or device study
14. Unwilling or unable to comply with the protocol or follow-up requirements
15. Any concurrent medical, psychological, or social condition, which may significantly interfere with the subject's optimal participation in the study, in the opinion of the investigator
16. Female patients of child-bearing potential.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2021-06-21 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
CTO Crossing | 12 months
  Successful crossing of the targeted chronic total occlusion, defined as angiography confirmed guidewire placement in the true lumen without utilization of a re-entry device.

SECONDARY OUTCOMES:
CapBuster system safety from perforations | 12 months
  Freedom from CapBuster System related clinically significant perforations that require intervention
CapBuster system safety from embolizations | 12 months
  Freedom from CapBuster System related clinically significant embolizations that require intervention
CapBuster system safety from dissections | 12 months
  Freedom from CapBuster System related clinically significant flow-limiting (type C, D, E) dissections that require intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Jihad Mustapha, Dr, Principal Investigator — Advanced Cardiac & Vascular Centers for Amputation Prevention Grand Rapids, MI 49525 USA
Locations (1):
- St Antonius Ziekenhuis, Koekoekslaan 1, 3435 CM, Nieuwegein, Netherlands

IPD SHARING:
Plan to Share IPD: No